CLINICAL TRIAL: NCT00041301
Title: An International Field Study Of The Reliability And Validity Of The EORTC QLQ-C30 And A Disease-Specific Questionnaire Module (QLQ-PR25) For Assessing Quality Of Life Of Patients With Prostate Cancer
Brief Title: Assessing Quality of Life of Patients With Prostate Cancer
Status: Completed | Type: Observational
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Other Study IDs: EORTC-15011-30011; EORTC-15011 (Other: EORTC); EORTC-30011 (Other: EORTC)
Record Dates: First submitted 2002-07-08; First posted 2003-01-27 (Estimated); Last update posted 2012-08-27 (Estimated); Status verified 2012-08

CONDITIONS: Prostate Cancer
Keywords: stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- QoL in prostate cancer: The study sample will be composed of a consecutive series of prostate cancer patients, stratified by stage of disease, local and locally advanced versus advanced (metastatic) disease, and undergoing active anti-tumor therapy. In order to increase sample homogeneity, and to facilitate evaluation of the responsiveness of the quality of life instruments to changes in patients' health status and symptoms experience over time, the subsample of patients with local or locally advanced disease will be restricted to those undergoing surgery (radical prostatectomy) or radiation therapy, and the subsample of metastatic disease patients will be limited to those receiving hormonal therapy.
  Interventions: Other: QoL assessment

INTERVENTIONS:
Other: QoL assessment — qol questionnaires
  Other Names: QLQ-C30; QLQ-PR25

SUMMARY:
RATIONALE: Quality of life assessment in patients undergoing prostate cancer treatment may help determine the intermediate and long-term effects of the treatment on these patients.

PURPOSE: Clinical trial to study the effectiveness of two questionnaires in assessing quality of life of patients who have prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess the scale structure, psychometric validity, and reliability of quality of life measurements using the EORTC QLQ-C30 and the prostate cancer-specific QLQ-PR25 questionnaires in patients with stage I-IV prostate cancer.

OUTLINE: This is a multicenter study. Patients are stratified according to stage of disease (local or locally advanced disease vs metastatic disease).

Patients complete EORTC QLQ-C30 and prostate cancer-specific QLQ-PR25 questionnaires before therapy and at 3 months after the start of therapy. Patients in stratum II also complete questionnaires at 6 months after the start of therapy.

PROJECTED ACCRUAL: A total of 375 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed prostate cancer
* Stratum I:

  * Clinically localized primary prostate cancer

    * T1-T3, G1-G3, N0, M0
    * Plan to undergo a radical prostatectomy OR
  * Local or locally advanced primary prostate cancer

    * T1-T4, G1-G3, N0, M0
    * Plan to undergo radiotherapy with curative intent
* Stratum II:

  * Metastatic prostate cancer

    * T1-T4, G1-G3, N1, M0-M1 OR
    * T1-T4, G1-G3, N0-1, M1
    * Plan to receive hormonal treatment

      * No anti-androgen monotherapy
* No cerebral metastases

PATIENT CHARACTERISTICS:

Age:

* Any age

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* Mentally fit to complete a questionnaire
* Literate in the language of the questionnaires
* No psychological, familial, sociological, or geographical condition that would preclude compliance
* No other concurrent malignancy except basal cell skin cancer
* No concurrent participation in other quality of life investigations that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* See Disease Characteristics
* No prior neoadjuvant hormonal treatment
* Planned adjuvant hormonal therapy (orchiectomy, luteinizing hormone-releasing hormone analogue, or maximal androgen blockade) is allowed for patients in stratum I

Radiotherapy:

* See Disease Characteristics
* No interstitial radiotherapy
* More than 2 years since prior radiotherapy (stratum II)

Surgery:

* See Disease Characteristics
* More than 2 years since prior prostatectomy (stratum II)

Other:

* No prior treatment for prostate carcinoma

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prostate cancer
Sampling Method: Non-Probability Sample
Enrollment: 625 (Actual)
Dates: Start 2002-03; Primary Completion 2004-12 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
psychometric validity of the PR25 module | before start of treatment, three months after the start of primary treatment and six months after the start of primary treatment.
  Quality of life scores will be evaluated for psychometric validity by:
  * Scale structure using multi-trait scaling analysis
  * Reliability using tests of internal consistency
  * Test-retest reliability
  * Validity using inter-scale correlations and known group comparisons
  * Sensitivity to change using two measurements of Quality of Life and ANOVA to look for the significance of changes in quality of life scores as a function of observed changes in clinical status over time.

SECONDARY OUTCOMES:
debriefing questionnaire information | at baseline
  Patients will be asked to complete a short debriefing questionnaire covering questions about the time taken to complete the EORTC QLQ-C30 and QLQ-PR25; the need for help in completing the questionnaires and querying whether any of the questionnaire items were confusing; difficult to answer or upsetting.

CONTACTS AND LOCATIONS:
Overall Officials: Neil K. Aaronson, PhD, Study Chair — The Netherlands Cancer Institute; George Van Andel, MD, Principal Investigator — Onze Lieve Vrouwe Gasthuis
Locations (33):
- Sir Charles Gairdner Hospital - Perth, Perth, Western Australia, Australia
- Belgium (6):
  - Academisch Ziekenhuis der Vrije Universiteit Brussel, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - Virga Jesse Hospital, Hasselt
  - Cazk Groeninghe - Campus Maria's Voorzienigheid, Kortrijk
  - U.Z. Gasthuisberg, Leuven
- Rigshospitalet, Copenhagen, Denmark
- Hopital Jean Bernard, Poitiers, France
- Germany (2):
  - Universitaetsklinikum Bonn, Bonn
  - Universitaets-Krankenhaus Eppendorf, Hamburg
- Italy (5):
  - Spedali Civili, Brescia
  - Istituto Scientifico H. San Raffaele, Milan
  - Azienda Ospedaliera Maggiore Della Carita, Novara
  - Universita di Palermo, Palermo
  - Azienda Sanitaria Ospedale San Giovanni Battista Molinette di Torino, Torino
- Netherlands (9):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Academisch Medisch Centrum, Amsterdam
  - Rijnstate Hospital, Arnhem
  - Academisch Ziekenhuis Groningen, Groningen
  - University Medical Center Nijmegen, Nijmegen
  - University Medical Center Rotterdam at Erasmus Medical Center, Rotterdam
  - Daniel Den Hoed Cancer Center at Erasmus Medical Center, Rotterdam
  - St. Elisabeth Ziekenhuis, Tilburg
- Norwegian Radium Hospital, Oslo, Norway
- Romania (2):
  - Inselspital, Bern, Bucharest
  - Institute of Oncology - Bucarest, Bucharest
- Turkey (Türkiye) (2):
  - Marmara University Hospital, Istanbul
  - Dokuz Eylul University School of Medicine, Izmir
- United Kingdom (3):
  - Bristol Haematology and Oncology Centre, Bristol, England
  - Velindre Cancer Center at Velinde Hospital, Cardiff, Wales
  - University of Wales College of Medicine, Cardiff, Wales

REFERENCES:
- [Result] Arraras JI, Villafranca E, Arias de la Vega F, Romero P, Rico M, Vila M, Asin G, Chicata V, Dominguez MA, Lainez N, Manterola A, Martinez E, Martinez M. The EORTC Quality of Life Questionnaire for patients with prostate cancer: EORTC QLQ-PR25. Validation study for Spanish patients. Clin Transl Oncol. 2009 Mar;11(3):160-4. doi: 10.1007/s12094-009-0332-z. PMID 19293053
- [Result] Arraras Urdaniz JI, Villafranca Iturre E, Arias de la Vega F, Dominguez Dominguez MA, Lainez Milagro N, Manterola Burgaleta A, Martinez Lopez E, Romero Rojano P, Martinez Aguillo M. The eortc quality of life questionnaire QLQ-C30 (version 3.0). Validation study for Spanish prostate cancer patients. Arch Esp Urol. 2008 Oct;61(8):949-54. doi: 10.4321/s0004-06142008000800017. PMID 19040169